CLINICAL TRIAL: NCT00291655
Title: A Multicenter, Open-label, Follow-up Trial Evaluating the Long-term Safety of Levetiracetam, for Patients Suffering From Epilepsy and Coming From the Study N01175 (NCT00175903).
Brief Title: Follow up Trial for Keppra (Levetiracetam) as Monotherapy in Patients With Newly Diagnosed Epilepsy Coming From N01175 (NCT00175903).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01237; EUDRACT NUMBER: 2006-000173-29
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Epilepsy
Keywords: NEWLY DIAGNOSED EPILEPSY; LEVETIRACETAM; KEPPRA; N01175 (NCT00175903)
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (LEV) (Experimental)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — 500 mg oral tablets,1000 - 3000 mg/day, twice a day (BID), duration of the study

SUMMARY:
For ethical reasons to give opportunity for adult subjects (≥16 or 18 years) suffering from newly diagnosed epilepsy who completed the therapeutic confirmatory, open-label trial N01175 (NCT00175903) conducted with levetiracetam in monotherapy and who benefited from the treatment, to receive treatment with levetiracetam until the monotherapy indication for levetiracetam is granted in Europe.

To continue to assess safety of levetiracetam as per adverse event reporting and observation of weight changes.

ELIGIBILITY:
Inclusion Criteria:

* Male/female adult subjects (≥ 16 or 18 years)
* Diagnosis of epilepsy (all types of seizures may be included)
* Subjects who completed N01175 (NCT00175903) trial and benefited from levetiracetam monotherapy

Other inclusion criteria may apply

Exclusion Criteria:

* Subjects withdrawn from N01175 (NCT00175903) trial for any reason
* Subjects who received treatment other than levetiracetam in N01175 (NCT00175903) trial
* Subject requiring add-on antiepileptic treatment
* Subjects from countries where levetiracetam is authorized for use as monotherapy in epilepsy treatment
* Sexually active woman with childbearing potential who is not using a medically accepted birth control method

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (35):
- Belgium (8):
  - Bruges
  - Edegem
  - Ghent
  - Haine-Saint-Paul
  - Jette
  - Kortrijk
  - Leuven
  - Ostend
- Bulgaria (2):
  - Sofia
  - Varna
- Finland (3):
  - Hus (helsinki)
  - Kuopio
  - Tampere
- France (13):
  - Blaye
  - Bordeaux
  - Brest
  - Carcassonne
  - Cherbourg
  - Lille
  - Lyon
  - Nancy
  - Rennes
  - Saint-Brieuc
  - Saint-Quentin
  - Toulouse
  - Valenciennes
- Poland (5):
  - Częstochowa
  - Krakow
  - Olsztyn
  - Poznan
  - Warsaw
- Switzerland (4):
  - Biel
  - Lausanne
  - Sankt Gallen
  - Zurich

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants Flow describes all subjects treated at least once during open-label monotherapy with Levetiracetam.
Groups:
- Levetiracetam Open- Label Treatment: Open-label treatment with Levetiracetam 500 mg oral tablets in monotherapy, 1000 - 3000 mg/day bid over up to 18 months
Period: Overall Study
Arm/Group | Levetiracetam Open- Label Treatment
Started | 130
Completed | 115
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam Open- Label Treatment
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.68 (18.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 72
Region of Enrollment [Number; unit: participants]
  France | 18
  Finland | 9
  Poland | 32
  Belgium | 25
  Bulgaria | 31
  Switzerland | 15

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Safety of Levetiracetam as Per Adverse Event (AE) Reporting in Open-label Therapy Phase
Description: Summarization for occurrence of adverse events like number of subjects with any adverse events or drug related adverse events is provided (see categories).
Time Frame: during open-label therapy phase of 18 months
Population: Safety population that includes all subjects that have been treated once.
Measure: Number; unit: participants
Arm/Group | Levetiracetam Open- Label Treatment
Number analyzed (Participants) | 130
participants
  Subjects with at least one AE | 40
  Subjects with AEs leading to dose change | 8
  Subjects with AEs leading to trial discontinuation | 1
  Subjects with drug-related AEs | 16
  Subjects with AEs of severe intensity | 4
  Subjects with serious AEs | 6
  Subjects with study drug-related serious AEs | 0
  Number of deaths | 0

2. Secondary Outcome: Change From Baseline in Body Weight to Withdrawal or End of Study After 18 Months
Time Frame: Start of open-label therapy (Baseline) to withdrawal or end of study after 18 months
Population: Subjects with a discontinuation visit
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Levetiracetam Open- Label Treatment
Number analyzed (Participants) | 79
kg | 0.71 (3.16)

ADVERSE EVENTS:
Time Frame: Open-label treatment over 18 months
Arm/Group | Levetiracetam Open- Label Treatment
Serious Adverse Events (participants affected / at risk) | 6/130
Other Adverse Events (participants affected / at risk) | 10/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam Open- Label Treatment (N=130)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam Open- Label Treatment (N=130)
Weight decreased (Investigations) | 3 (3)
Weight increased (Investigations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.